CLINICAL TRIAL: NCT00686660
Title: A Multi-Center Study of Rehabilitation to Stable Chronic Obstructive Pulmonary Disease (COPD) Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Chao Yang Hospital (Other)
Collaborators: Beijing Tongren Hospital (Other); Xuanwu Hospital, Beijing (Other); Beijing Fuxing Hospital (Unknown); Peking University First Hospital (Other); Beijing Miner General Hospital (Unknown); Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other); Beijing Shuyi Hospital (Other); Beijing Daxing Hospital (Unknown); Beijing Huairou Hospital (Other)
Responsible Party: chen wang, beijing chaoyang hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COPD rehabilitation CYH 2007
Record Dates: First submitted 2008-05-27; First posted 2008-05-30 (Estimated); Last update posted 2008-06-17 (Estimated); Status verified 2008-05

CONDITIONS: COPD; Inflammation
Keywords: copd; rehabilitation; quality of life; inflammation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Inflammation | interventions — Walking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): C-W G: in training period, patients do cycling on cycle ergometry at hospital. in non-training period, patients walk at community.
  Interventions: Behavioral: cycling, walking
- 2 (Other): C-nonW G: in training period, patients do cycling at cycle ergometry at hospital, in non-training period, patients don't walk at community.
  Interventions: Behavioral: cycling, non-walking
- 3 (Experimental): W-W G: in training period, patients do walking along 60 meters place at hospital, in non-training period, patients do walking in community
  Interventions: Behavioral: walking, walking
- 4 (Other): W-nonW G: in training period, patients do walking along 60 meter place, in non-training period,patients don't walk at community.
  Interventions: Behavioral: walking, non-walking

INTERVENTIONS:
Behavioral: cycling, walking — In training period, patients do cycling on cycle ergometry. two times per week, 8 weeks per training period, two training period per year, two years.
  In non-training period, patients do walking at community. four days per week,18 weeks per non-training period, two non-training period per year, two years.
  Other Names: no.
  Arms: 1
Behavioral: cycling, non-walking — In training period, patients do cycling. two times a week, 8 weeks per training period, two training period per year, two years.
  In non-training period, patients don't receive walk training.
  Other Names: no.
  Arms: 2
Behavioral: walking, walking — In training period, patients do walking at hospital, two times per week, 8 weeks per training period, two training period per year, two years.
  In non-training period, patients do walking at community, four days per week, 18 weeks per non-training period, two non-training period per year, two years.
  Other Names: no.
  Arms: 3
Behavioral: walking, non-walking — In training period, patients do walking at hospital, two times per week, 8 weeks per training period, two training period per year, two years.
  In non-training period, patients don't walking at community.
  Other Names: no.
  Arms: 4

SUMMARY:
This is a multi-center prospective follow-up study.

* to choose the stable COPD patients in community
* to compare different modes of exercise (cycling and walking)
* to compare the effect of different exercises on the quality of life,exercise endurance,dyspnea and depression

DETAILED DESCRIPTION:
This is a multi-center prospective follow-up study.More than 20 hospitals participate the research. More than 300 stable COPD patients will be recruited.It is a two-year study. There are four groups, cycling and walking group(C-WG),cycling and non-walking group(C-nonWG),walking and walking group(W-WG),walking and non-walking group(W-nonWG).

1. All patients from four groups will finish baseline investigation and blood sample, including informed consent,questionaires(SGRQ,CRDQ,MRCQ,Depression Scale,etc.),spirometry,6MWT,MIP,MEP,BMI,CRP,TNF,IL-8, etc.Patients in C-WG and C-nonWG will finish cardiopulmonary test.
2. Patients receive 8 weeks training program, includes upper and lower extremities endurance exercises and respiratory muscle endurance exercises. Patients in both CGs cycling at cycle ergometry. Patients in W-WG and W-nonWG walking instead. All patients receive training program twice per year, for two years. Patients were supervised by physicians or nurses at hospital while they are training.
3. In the non-training period, patients in W-WG and C-WG will continue to walk at community, supervised by nurses who call them every month. The other two groups(C-nonWG and W-nonWG) do not receive special requirement on exercise.
4. Telephone call interview will give to patients every month to find whether they have acute exacerbation. Patients are asked to record their activities during daytime in the diary cards.
5. All patients will finish investigation and blood sample after one year and two year,including questionaires,spirometry,6MWT,MIP,MEP,BMI,CRP,TNF,IL-8, etc.Patients in CG will finish cardiopulmonary test.

ELIGIBILITY:
Inclusion Criteria:

* according to GOLD, patients who are diagnosed as COPD, lung function at II or III grades (II:50%≤FEV1<60%pre；III:30%≤FEV1<50%pre）；
* 40≤age≤75 years old；
* don't have acute exacerbation in the past one month；
* SpO2 > 88% at rest；

Exclusion Criteria:

* diabetes,blood glucose don't control well;
* vascular diseases(vasculitis,deep venous thrombosis,varicose veins, etc);
* joint diseases which may affect activities;
* cerebrovascular diseases which may affect activities;
* unstable angina during the past 1 month of acute myocardial infarction in the past 6 months;
* severe arrhythmia;
* cardia insufficiency;
* hypertension which don't control well(systolic pressure>160mmHg and/or diastolic pressure> 100mmHg);
* chronic liver or renal insufficiency;
* cognitive handicap.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2007-09; Primary Completion 2010-06 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
quality of life, dyspnea score, exercise endurance, depression,markers of inflammation (CRP, TNF, IL-8) | two years

CONTACTS AND LOCATIONS:
Overall Officials: chen wang, phD, Principal Investigator — Beijing Chao Yang Hospital
Locations (1):
- Beijing Chaoyang Hospital, Beijing, Beijing Municipality, China